CLINICAL TRIAL: NCT06764095
Title: CAST-AI: Cystectomy After Systemic Therapy With ADC and Immunotherapy
Brief Title: Enfortumab Vedotin and Pembrolizumab With Cystectomy and/or Ureterectomy for Locally Advanced or Metastatic Bladder and Upper Urothelial Tract Cancer, CAST-AI Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240504; NCI-2024-10405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006857 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-12-27; First posted 2025-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Bladder Urothelial Carcinoma; Locally Advanced Renal Pelvis and Ureter Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis and Ureter Urothelial Carcinoma; Stage III Bladder Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis and Ureter Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms | interventions — Specimen Handling; Cystectomy; enfortumab vedotin; Hyperthermia, Induced; Magnetic Resonance Spectroscopy; pembrolizumab; Nephroureterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (enfortumab vedotin, pembrolizumab) (Experimental): Patients receive standard of care enfortumab vedotin IV over 30 minutes on day 1 and day 8 and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for at least 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity. Patients who are surgical candidates may then undergo cytoreductive cystectomy and/or ureterectomy. Patients may also undergo MDT at any time per standard of care. After surgery, patients may then continue to receive maintenance enfortumab vedotin and pembrolizumab. Additionally, patients undergo urine and blood sample collection, CT, PET/CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystectomy; Drug: Enfortumab Vedotin; Procedure: Local Therapy; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Ureterectomy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Cystectomy — Undergo cytoreductive cystectomy
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG 22CE; ASG-22CE; ASG22CE; Enfortumab Vedotin-ejfv; Padcev
Procedure: Local Therapy — Undergo MDT
  Other Names: Localized Therapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; QL2107; RPH 075; RPH-075; RPH075; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Ureterectomy — Undergo ureterectomy

SUMMARY:
This phase IV trial tests the impact of standard of care enfortumab vedotin and pembrolizumab followed by removal of all or part of the bladder (cytoreductive cystectomy) and/or removal of all or part of the tube that carriers urine from the kidneys to the bladder (ureterectomy) on outcomes in patients with bladder and upper urothelial tract that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of tumor cells. Enfortumab attaches to a protein called nectin-4 on tumor cells in a targeted way and delivers vedotin to kill them. It is a type of antibody-drug conjugate. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor and may interfere with the ability of tumor cells to grow and spread. Giving standard of care enfortumab vedotin and pembrolizumab followed by cytoreductive cystectomy and/or ureterectomy (CC/U) may improve outcomes in patients with locally advanced or metastatic bladder or upper urothelial tract cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate progression-free survival at 12 months in patients undergoing treatment with enfortumab vedotin and pembrolizumab (EV/Pembro) and CC/U with or without metastasis-directed therapy (MDT).

SECONDARY OBJECTIVES:

I. To evaluate overall response rate (ORR). II. To evaluate surgical candidacy rate (defined as the proportion of patients in the study who undergo cystectomy and/or ureterectomy) and pathologic complete response and downstaging (ypT0, ypTis/Ta) at time of CC/U.

III. To evaluate progression-free survival (PFS). IV. To evaluate overall survival (OS). V. To evaluate the toxicity profile as assessed per Common Terminology Criteria for Adverse Events (CTCAE).

CORRELATIVE OBJECTIVES:

I. Determine the prognostic value of exosomes and circulating cell-free deoxyribonucleic acid (cfDNA) minimal residual disease (MRD) markers.

II. Determine the prognostic value of exosomes and cfDNA as early indicators of disease relapse.

III. Characterize duration of response. IV. Evaluate treatment tolerability as assessed per Patient Reported Outcomes (PRO) (CIPN20).

OUTLINE:

Patients receive standard of care enfortumab vedotin intravenously (IV) over 30 minutes on day 1 and day 8 and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for at least 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity. Patients who are surgical candidates may then undergo cytoreductive cystectomy and/or ureterectomy. Patients may also undergo MDT at any time per standard of care. After surgery, patients may then continue to receive maintenance enfortumab vedotin and pembrolizumab. Additionally, patients undergo urine and blood sample collection, computed tomography (CT), positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up every 9 weeks for up to 18 months, then every 12 weeks up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of informed consent
* Histologically proven urothelial carcinoma [American Joint Committee on Cancer (AJCC) 2017] of the bladder (BCa) or upper urothelial tract (UTUC), N+ and/or M+. Initial diagnosis must be within 90 days of planned date for treatment initiation

  * The following variant histologic subtypes are permitted in any amount

    * Urothelial with squamous differentiation
    * Urothelial with sarcomatoid differentiation
  * Mixed variant histologic subtypes are permitted if urothelial differentiation is predominant (e.g., < 50% variant histologic subtype)
* Willing to undergo cytoreductive cystectomy (CC) or ureterectomy (U) and deemed clinically a surgical candidate (presuming good response) by the attending urologist
* Eastern Cooperative Oncology Group (ECOG) performance status grade 0, 1, or 2
* Hemoglobin ≥ 8.0 g/dL (obtained ≤ 28 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 28 days prior to registration)
* Platelet count ≥ 80,000/mm^3 (obtained ≤ 28 days prior to registration)
* Alanine aminotransferase (ALT) OR aspartate transaminase (AST) ≤ 3.5 x upper limit of normal (ULN) (obtained ≤ 28 days prior to registration)
* Total bilirubin ≤ 3 x ULN OR direct bilirubin ≤ 3 x ULN (obtained ≤ 28 days prior to registration)
* Estimated glomerular filtration rate ≥ 15 ml/min (obtained ≤ 28 days prior to registration)
* Prior systemic chemotherapy for indications other than urothelial cell carcinoma of the bladder is permitted, but interval between this treatment and study enrollment must exceed 24 months
* All adverse events associated with any prior surgery must have resolved to CTCAE version 5.0 grade < 2 prior to registration
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study and agree to store samples when applicable
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* The following histologic variants/divergent differentiation are excluded from trial participation:

  * Presence of urothelial carcinoma with histologic variants comprising > 50% of histology
  * Any amount: neuroendocrine, micropapillary, or signet ring cell features
* Prior systemic chemotherapy for urothelial cell carcinoma of the bladder at any time (excluding intravesicular therapies)
* Known active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are:

  * Skin cancer (non-melanoma or melanoma) that is considered completely cured
  * Non-invasive cervical cancer treated that is considered completely cured
  * Breast cancer:

    * Adequately treated lobular carcinoma in situ or ductal carcinoma in situ considered to have a very low risk of recurrence
  * Localized prostate cancer (T1c/T2N0M0):

    * Gleason score 6, treated by either surgery or ablation within the last 24 months or untreated and under active surveillance
    * Gleason score 3+4 that has been treated (may include surgery or ablation) within the last 24 months and considered to have a very low risk of recurrence (i.e., cT1c or pT2 on prostatectomy specimen)
* Received prior systemic chemotherapy or targeted small molecule therapy (excluding hormonal therapy) within 2 years prior to starting study treatment
* History of uncontrolled adrenal insufficiency
* History of uncontrolled cardiovascular disease including any of the following in the preceding 6 months: unstable angina, myocardial infarction, ventricular fibrillation, Torsades de Pointes, cardiac arrest, or known congestive New York Heart Association class III-IV heart failure, cerebrovascular accident, or transient ischemic attack; pulmonary embolism or other venous thromboembolism
* Known active tuberculosis
* Is receiving immunosuppression for an allogeneic tissue/solid organ transplant
* Participants with an active autoimmune disease requiring systemic treatment. Participants with autoimmune disorders not requiring systemic treatment (eg, skin conditions such as vitiligo or alopecia) or conditions requiring hormonal replacement therapies such as type 1 diabetes mellitus or hypothyroidism are permitted to enroll
* Known clinically significant liver disease that precludes participant treatment regimens prescribed on the study (including, but not limited to active viral, alcoholic, or other autoimmune hepatitis, cirrhosis, or inherited liver disease)
* Known human immunodeficiency virus (HIV) infection, unless the participant has been on a stable antiretroviral therapy regimen for the last 6 months or more and has had no opportunistic infections and a CD4 count of > 350 in the last 6 months
* Known active hepatitis B or C infection [however, participants with history of hepatitis C infection but normal hepatitis C virus polymerase chain reaction test and participants with hepatitis B with positive hepatitis B surface antigen (HBsAg) antibody are allowed]
* Known urinary tract infection (UTI), defined as a symptomatic infection with a positive urine culture with a bacterial count of ≥ 10^5 colony forming units (CFU)/mL in urine voided from women, or > 104 CFU/mL in urine voided from men, or in straight catheter urine from women. Symptoms may include dysuria, urgency, frequency, and/or systemic symptoms such as fever, chills, elevated white blood cell, and/or abdominal/flank pain. Participants free from symptoms for 7 days with no culture evidence of ≥ 10^5 CFUs may be eligible
* Known active, uncontrolled urogenital bacterial, viral or fungal infections, including UTI. Skin/nail fungal infections are not exclusionary. Participants with active shingles (varicella zoster infection) will be excluded from the study
* Evidence of interstitial lung disease or active non-infectious pneumonitis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants who have had a history of acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation
* Known history of impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions
* Pelvic radiotherapy administered at any time
* Received a live virus vaccine within 30 days of planned start of study treatment
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Active infection requiring systemic intravenous therapy within 30 days prior to planned treatment initiation
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Participants with a history of grade ≥ 3 toxic effects when using anti-tumor necrosis factor (TNF) or anti-interleukin (IL)-6 agents are excluded
* Participants still recovering from toxicity of prior anticancer therapy which was received more than 24 months prior to enrollment (except toxicities which are not clinically significant such as alopecia, skin discoloration)
* Participants who require immunosuppressive medications including but not limited to systemic corticosteroid at doses > 10 mg/day of prednisone or its equivalence, methotrexate, cyclosporine, azathioprine, and TNF alpha blockers. Use of immunosuppressive medications for the management of immune related adverse events, infusion related reactions, or in participants with contrast allergies is acceptable. Use of inhaled, topical, and intranasal corticosteroids are permitted
* Participants with a history of allergy to protein-based therapies and participants with a history of any significant drug allergy (such as anaphylaxis, hepatotoxicity, or immune mediated thrombocytopenia or anemia) are excluded
* Currently participating or has participated in a study of an investigational agent and received study therapy or investigational device within 4 weeks prior to enrollment
* Participants who have not recovered from the effects of major surgery or significant traumatic injury at least 14 days before registration [transurethral resection of bladder tumor (TURBT) is not considered major surgery]. Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participants (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* The participant is unable to comply with the requirements of this protocol, including any factors that are likely to affect the participant's return for scheduled visits and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 12 months | At 12 months
  Will be calculated as the number of patients who are alive and progression-free at 12 months after study enrollment. Progression will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria.

SECONDARY OUTCOMES:
PFS overall | Up to 5 years
  PFS will be defined as the time from study registration to the date of death due to any cause or progressing disease, whichever occurs first. Progression will be determined by RECIST v1.1 criteria.
Overall survival (OS) | Up to 5 years
  OS will be defined as time from the date of registration to the date of death from any cause
Overall response rate (ORR) | Up to 5 years
  ORR will be defined as confirmed complete response (CR) or partial response (PR) according to RECIST v 1.1 criteria, assessed at the time of cytoreductive cystectomy and/or ureterectomy (CC/U) or at time of best response during treatment.
Surgical candidacy rate | Up to 5 years
  Will be defined as the proportion of patients in the Modified Intent-to-Treat (mITT) population who undergo CC/U [cytoreductive cystectomy (CC) and/or ureterectomy (U)].
Pathologic complete response (pCR) rate | Up to 5 years
  Will be defined defined as the absence of viable tumor cells in the cystectomy. The pCR rate will be estimated as the number of patients experiencing a pCR.
Downstaging | Baseline (at time of CC/U)
  Assessed as the number of patients achieving downstaging (ypT0, ypTis/Ta) at the time of CC/U.
Incidence of adverse events (AEs) | Up to 18 months after cycle 1 day 1 (C1D1); cycle length = 3 weeks
  The maximum grade for each type of AEs will be recorded for each patient. Frequency tables will be reviewed to determine patterns. The rate of patients experiencing at least one grade 3+, 4+, or 5 adverse event (regardless of attribution) will be reported.
Patient-reported quality of life | Up to 18 months after cycle 1 day 1 (C1D1); cycle length = 3 weeks
  Patient-reported quality of life will be assessed according to the Chemotherapy-Induced Peripheral Neuropathy (CIPN20). The mean CIPN20 total score will be reported at each of the protocol-defined timepoints, and mean patient-level changes from baseline total score will also be reported at each of the post-baseline protocol-defined timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J. Orme, MD, PhD, Principal Investigator — Mayo Clinic in Rochester; Paras H. Shah, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials